CLINICAL TRIAL: NCT05642195
Title: Phase I/II Evaluation of a Cancer Lysate Vaccine and Montanide(R) ISA-51 VG With or Without the IL-15 Super-Agonist N-803 as Adjuvant Therapy for PD-L1 Negative Non-Small Cell Lung Cancer
Brief Title: Evaluation of a Cancer Lysate Vaccine and Montanide (Registered Trademark) ISA-51 VG With or Without the IL-15 Super-Agonist N-803 as Adjuvant Therapy for PD-L1 Negative Non-Small Cell Lung Cancer
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Revisions to eligibility/design being made prior to enrollment of first participants.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 10000520; 000520-C
Record Dates: First submitted 2022-12-06; First posted 2022-12-08 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-07-28

CONDITIONS: Non-Small Cell Lung Cancer; Non-Small Cell Lung Carcinoma; Carcinoma, Non-Small-Cell Lung; Carcinomas
Keywords: Immunotherapy; NSCLC; H1299 Cell Lysates; No Clinical Evidence Of Active Disease (Ned); Minimal Residual Disease (Mrd); Disease-Free Survival (Dfs); Ct-X Antigens; Autosomal Ct Antigens; Cell Mediated Response
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma; Neoplasm, Residual | interventions — Monatide (IMS 3015); ALT-803; Biological Assay

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1/ Vaccine with Montanide Adjuvant (Experimental): H1299 cell lysate vaccine administered with Montanide (Registered Trademark) ISA-51 VG adjuvant without or with N-803 (Phase I component to determine H1299 cell lysate dose)
  Interventions: Biological: Montanide (Registered Trademark) ISA-51 VG Adjuvant; Biological: H1299 Cell Lysates; Drug: N-803; Device: Ventana PD-L1 (SP263 or SP142) assay
- 2/ Vaccine with Montanide Adjuvant and N-803 (Experimental): H1299 cell lysate vaccine administered with Montanide (Registered Trademark) ISA-51 VG adjuvant with N-803 (H1299 cell lysate at dose determined in Phase I)
  Interventions: Biological: Montanide (Registered Trademark) ISA-51 VG Adjuvant; Biological: H1299 Cell Lysates; Drug: N-803; Device: Ventana PD-L1 (SP263 or SP142) assay

INTERVENTIONS:
Biological: Montanide (Registered Trademark) ISA-51 VG Adjuvant — H1299 cell lysate with Montanide (Registered Trademark) ISA-51 VG adjuvant vaccine via subcutaneous injections once every cycle (1 cycle=28 days) for 6 cycles (i.e., 6 vaccinations). Dose Level 1 (DL1) starting dose is 20 mcg lysate protein in 2-2.5 mL Montanide (Registered) ISA-51 VG adjuvant; lysate concentration will be 8-10 mcg/mL. Additional 2 vaccine injections for subjects with immunologic response and NED.
Biological: H1299 Cell Lysates — H1299 cell lysate with Montanide (Registered) ISA-51 VG adjuvant vaccine via subcutaneous injections once every cycle (1 cycle=28 days) for 6 cycles (i.e., 6 vaccinations). Dose Level 1 (DL1) starting dose is 20 mcg lysate protein in 2-2.5 mL Montanide (Registered Trademark) ISA-51 VG adjuvant; lysate concentration will be 8-10 mcg/mL. Additional 2 vaccine injections for subjects with immunologic response and NED.
Drug: N-803 — N-803 via subcutaneous injection in the abdomen at dose of 15 ug/kg every 4 weeks, on Day 1 of each cycle. N-803 dosing will be calculated using a weight obtained within 5 days prior to the first dose. Dose re-calculated at the beginning of each subsequent cycle in the event of a 10% or greater weight change.
Device: Ventana PD-L1 (SP263 or SP142) assay — FDA-approved assays used off-label for study as treatment determining in-vitro diagnostic devices to assess subject PD-L1 quantitation. Testing will be performed on provided archival samples or on fresh sample that is collected at screening for confirmation of diagnosis; no additional sample collection for purposes of PD-L1 testing.

SUMMARY:
Background:

Surgery is the primary treatment for non-small cell lung cancer (NSCLC) that is diagnosed in its earlier stages. But the tumors often return. Radiation and chemotherapy can improve survival in some people who have had surgery for NSCLC, but these treatments also cause serious side effects. A new approach, called immunotherapy, may be a better way to stop NSCLC tumors from coming back.

Objective:

To test a new treatment (H1299 lung cancer cell vaccine combined with the drug N-803) in people who received surgery for NSCLC.

Eligibility:

Adults aged 18 years or older with no sign of disease after surgery for NSCLC.

Design:

Participants will be screened. They will have a physical exam with blood tests. They will have tests of their heart and lung function. They will have imaging scans.

Study treatment will be given in 28-day cycles. Participants will visit the clinic on the first day of each cycle. They will receive 2 treatments at each visit:

The study vaccine is given as 2-4 small shots under the skin of the thigh or arm.

N-803 is given as a shot under the skin of the abdomen.

Treatment will continue for 6 cycles. Blood tests and imaging scans will be repeated throughout the study.

Participants will have a blood test 1 month after receiving the 6th vaccine. Some participants may then resume taking N-803; they may also receive 2 more vaccinations at 3 and 6 months after their previous treatment.

Follow-up visits will continue for up to 5 years.

DETAILED DESCRIPTION:
Background:

* Cancer-testis (CT) antigens (CTA), particularly those encoded by genes on the X chromosome (CT-X antigens) have emerged as attractive targets for cancer immunotherapy.
* Recent studies suggest that CT-X antigens which are up regulated by epigenetic mechanisms may be preferentially expressed in pluripotent stem/tumor initiating cells that mediate treatment resistance and metastasis of human cancers.
* Whereas pulmonary malignancies express a variety of CT-X antigens, immune responses to these proteins are uncommon in lung cancer patients due to low-level, heterogeneous antigen expression, epigenetic repression of genes regulating antigen processing/presentation, and local as well as systemic immunosuppression in these individuals.
* Conceivably, vaccination of lung cancer patients with tumor cells expressing high levels of CT-X antigens in combination with regimens that inhibit immunosuppressive functions of T regulatory cells and enhance activity of natural killer (NK) cells will induce broad immunity to these antigens.

Primary Objectives:

* Phase I Component: To determine the safety of H1299 lung cancer cell lysate vaccines administered with Montanide (Registered Trademark) ISA-51 VG adjuvant and N-803.
* Phase II Component: To assess the frequency of immunologic responses to purified CT-X and autosomal CT antigens in NSCLC participants following vaccinations with H1299 cancer cell lysate and Montanide (Registered Trademark) ISA-51 VG adjuvant in combination with N-803.

Eligibility:

* Participants with pathologically confirmed Stage IB-IIIA (T2a-T4/N0, T1-T3N1, T1-T2/N2) NSCLC per 8th edition TNM Staging System non-small cell lung cancer (NSCLC) who have no clinical evidence of active disease (NED) following standard therapy completed within the past 12 weeks.
* Participants must be 18 years or older with an ECOG performance status of 0-2.
* Participants must have adequate bone marrow, kidney, liver, lung, and cardiac function.
* Participants receiving systemic immunosuppressive medications will be excluded.
* Participants with HIV will be excluded.

Design:

* Following recovery from surgery, and adjuvant therapy if indicated, eligible participants will be vaccinated via deep subcutaneous (SQ) injection with H1299 cell lysate and Montanide (Registered Trademark) ISA-51 VG (Trademark) adjuvant with or without subcutaneous N-803 monthly until six vaccinations have been given.
* Imaging studies will be performed at baseline, one month following the 3rd and 6th vaccinations, and at post-treatment follow-up (every 3 months for 3 years and then every 6 months for another 2 years, for 5 years total follow-up).
* Leukapheresis will be performed at baseline and at treatment evaluation one month following completion of the six vaccinations.
* Systemic toxicities and immunologic responses to therapy will be recorded.
* Pre- and post-vaccination serologic and cell mediated responses to a panel of CT-X antigens will be assessed before and one month following completion of the six vaccinations.
* Individuals deemed to have responded to vaccine treatment and exhibit no evidence of disease recurrence or secondary malignancy will be eligible for 2 additional vaccinations at 3 months after receiving the sixth vaccine and 6 months after receiving the 6th vaccine with N-803.
* Numbers and percentages of immune subsets, soluble factors, and cytokines in peripheral blood will be assessed before and after the six vaccinations.
* Immunologic responses to autologous tumor cells (if available) as well as pooled lung cancer stem cell vs. normal lung-induced pluripotent stem cell (Lu-iPSC) lysates will be evaluated in an exploratory manner.
* Up to 28 participants may receive study intervention on this protocol.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Participant with histologically or cytologically proven Stage IB-IIIA (T2a-T4/N0, T1- T3N1, T1-T2/N2) NSCLC per 8th edition TNM Staging System with no clinical evidence of active disease (NED) or minimal residual disease (MRD) not readily accessible by non-invasive biopsy or resection/radiation following standard therapy. Initial diagnosis must be confirmed by the NIH Laboratory of Pathology.
* History of PD-L1 expression in cancer cells < 1% as determined by IHC analysis.
* Participant must be enrolled within 12 weeks following completion of prior SOC therapy.
* Participant must have an ECOG performance status of 0-2.
* Participant must be >=18 years of age.
* Participant must be willing to co-enroll on protocol 06C0014 (Prospective Analysis of Genetic and Epigenetic Alterations in Patients with Thoracic Malignancies) allowing for the collection of blood for correlative experiments pertaining to this protocol and related translational research efforts in the Thoracic Surgery Branch.
* Participant must have evidence of adequate bone marrow reserve, hepatic and renal function as evidenced by the following laboratory parameters (all eligibility assessment/enrollment bloodwork must be done at NIH no more than 2 weeks prior to enrollment):
* Absolute neutrophil count greater than 1500/mm3
* Absolute lymphocyte count greater than 800/mm3
* Platelet count greater than 75,000/mm3
* Hemoglobin greater than 8 g/dL (participant may receive transfusions to meet this parameter)
* INR< 1.5xULN
* Total bilirubin < 1.5 x upper limits of normal (except those with Gilberts disease)
* Serum creatinine less than or equal to 1.6 mg/mL or the eGFR must be greater than 60 mL/min/1.73m2
* Seronegative for HIV antibody by bloodwork performed at NIH no more than 4 weeks prior to enrollment.
* Seronegative for active hepatitis B, and seronegative for hepatitis C antibody. If hepatitis C antibody test is positive, then patient must be tested for the presence of antigen by RTPCR and be HCV RNA negative by bloodwork performed at NIH no more than 4 weeks

prior to enrollment.

* Participants who are breastfeeding or plan to breastfeed must agree to discontinue/postpone breastfeeding while receiving investigational treatment and for 120 days after the last dose of vaccine or N-803.
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) within 28 days prior initiation of study therapy, for the duration of study participation and up to 120 days after the last

dose of the drug.

-Participant must be able to understand and willing to sign an informed consent.

EXCLUSION CRITERIA:

* Participants receiving other investigational agents.
* Participants on any active treatment for their cancer upon study entry.
* Participant who is initially rendered NED or have MRD following standard therapy but exhibit disease progression prior to initiation of vaccination.
* Participant requiring chronic systemic treatment with steroids above physiologic doses.
* Participant receiving warfarin anticoagulation, who cannot be transitioned to other agents such as enoxaparin or dabigatran, and for whom anticoagulants cannot be held for up to 24 hours.
* Participant with uncontrolled hypertension (> 160/95), unstable coronary disease evidenced by uncontrolled arrhythmias, unstable angina, decompensated CHF (> NYHA Class II), or myocardial infarction within 6 months prior to initiation of study therapy.
* Participant with any of the following pulmonary function abnormalities: FEV, < 35% predicted; DLCO < 35% predicted (post-bronchodilator); oxygen saturation less than 92% on room air based on assessment at NIH or outside medical facility no more than 4 weeks prior to protocol enrollment.
* Active COVID infection
* Participant pregnancy
* Uncontrolled intercurrent illness occurring within 3 months prior to initiation of study therapy /social situations (as assessed by social services) that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2033-12-30 (Estimated); Study Completion 2035-12-30 (Estimated)

PRIMARY OUTCOMES:
Phase II Component: To assess the frequency of immunologic responses to purified CT-X and autosomal CT antigens in NSCLC participants following vaccinations with H1299 cancer cell lysate and Montanide ISA-51 VG adjuvant in combination with N-803 | 1 month following first 6 vaccinations, and every 6 months during retreatment
  Analyses which investigate immunologic responses to a panel of CT antigens in vaccinated participants. Serologic response will be defined as new antibody reactivity to a CT antigen, increased titer of an existing antibody, or IgM-to-IgG class switch following vaccination. Cell Mediated response will be evaluated using Elispot or comparable assays.CT X antigen reactivity assessed by peripheral blood assays one month following the first six vaccinations, and every 6 months during retreatment.
Phase I Component: To determine the safety of H1299 lung cancer cell lysate vaccines administered with Montanide (Registered Trademark) ISA-51 VG adjuvant and N-803 | before each cycle, every 2 weeks between vaccines 1 & 2 (AE only), at each treatment evaluation, and at the safety visit
  Assessment of safety and tolerability of the lysate vaccine regimen (DL1 and/or DL-1) with N-803 as determined by the frequency and severity of adverse events: AEs assessed by laboratory evaluations (before each cycle, every 2 weeks between vaccines 1 & 2, at each treatment evaluation, and at the safety visit) and queries (before each cycle, at each treatment evaluation and at safety visit) from the start of study intervention through 30 days after the last dose of vaccine. Unsolicited AEs are assessed throughout the study including beyond safety visit.

SECONDARY OUTCOMES:
To determine disease-free survival (DFS) in lung cancer participants receiving adjuvant H1299 lung cancer cell lysate vaccines administered with Montanide (Registered Trademark) ISA-51 VG and N-803 | every 12 weeks while on treatment, during follow up for every 3 months for 3 years then every 6 months for 2 years or disease progression, final DFS evaluation visit
  Overall Survival (OS) and disease-free survival (DFS) determined from the on-study date until date of death, disease recurrence, loss of immune response, or last follow-up as appropriate using the Kaplan-Meier method. DFS by scans every 12 weeks while on treatment or continued treatment, and during follow up every 3 months for 3 years, every 6 months for another 2 years or through disease progression ending at time of final DFS evaluation for each participant at 5 years post enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: David S Schrump, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded will be shared upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data from this study may be requested from other researchers after the completion of the primary endpoint.
Access Criteria: Data from this study may be requested by contacting the PI.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_000520-C.html